CLINICAL TRIAL: NCT06585566
Title: Evaluation of Secondary Alveolar Cleft Reconstruction With Labial and Palatal Retromolar Cortical-Shells (A Case Series Study)
Brief Title: Alveolar Cleft Reconstruction With Cortical-Shells
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Amr Gibaly, Associate Professor of Oral and Maxillofacial Surgery, Beni-Suef University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Alveolar Cleft
Keywords: Bone graft; Cortical- shells; Radiographic Density; Horizontal bone gain; Vertical bone loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Secondary alveolar bone grafting (SBAG) (Other): A SABG technique that utilizes retromolar cortical shells and the underlying cancellous particulates to formulate a three-dimensional alveolar cleft reconstruction.
  Interventions: Procedure: Cortical-shell graft

INTERVENTIONS:
Procedure: Cortical-shell graft — Retromolar cortical shell graft technique for SABG

SUMMARY:
The main goal of the secondary alveolar bone grafting (SABG) for alveolar clefts is the rehabilitation of the disorganized maxilla, aiming to stabilize the maxillary foundation as a solid functional mass that would abort growth disturbance, allow for teeth eruption, and enhance their orthodontic movements.

The study evaluates the outcomes of a ( SABG) technique that utilizes the retromolar cortical shell technique to reconstruct the alveolar clefts.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes with an age range of (eight to fifteen years), with unilateral maxillary alveolar cleft.
2. good oral hygiene and general good health

Exclusion Criteria:

1. The evidence of clinical or radiographic signs of local maxillary pathosis or palatal fistulae.
2. Those patients with bilateral alveolar clefts, cleft-associated syndromes, and those with a systemic disease that would affect either bone harvest or graft healing.
3. A history of previous failed alveolar cleft reconstruction.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Horizontal bone width | 6 months consolidation period
  The amplitude of radiographic horizontal bone width change

SECONDARY OUTCOMES:
Vertical bone level | 6 months consolidation period
  The amplitude of radiographic vertical bone change
Bone density | 6 months consolidation period
  The radiographic bone density of the consolidated graft at the site of the reconstructed cleft

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Amr Gibaly, Cairo
  - Department of Oral and Maxillofacial Surgery, Faculty of Oral and Dental Medicine, Modern University for Technology & Information., Cairo

IPD SHARING:
Plan to Share IPD: No